CLINICAL TRIAL: NCT04103697
Title: A Multicenter Prospective Phase III Clinical Trial of Neoadjuvant CapOx Chemotherapy in Patients With Intermediate Risk Middle and Upper Rectal Cancer
Brief Title: Neoadjuvant Chemotherapy in Patients With Intermediate Risk Upper and Mid Rectal Cancer
Acronym: RuCorT-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Sergey Gordeyev, Principal Investigator, Consultant surgeon, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuCorT-01
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Rectal Neoplasms Malignant; Rectum Carcinoma; Rectal Cancer
Keywords: rectal cancer; neoadjuvant chemotherapy; mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4xCapOx (Experimental): Patients will receive 4 cycles of neoadjuvant CapOx chemotherapy (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 bid per os days 1-14 every 3 weeks). In case of partial response or stable disease (based on pelvic MRI) patients proceed to surgery. In case of disease progression patients receive 50 Gy pelvic chemoradiotherapy with capecitabine 825 mg/m2 bid per os on radiation days and then surgery. The decision to proceed with adjuvant chemotherapy postoperatively will be based on pTNM stage
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy; Procedure: Rectal cancer surgery
- Surgery (Active Comparator): Patients will receive standard surgery for rectal cancer with partial or total mesorectal excision (based on exact tumor location and surgeons discretion). The decision to proceed with adjuvant chemotherapy postoperatively will be based on pTNM stage
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Procedure: Rectal cancer surgery

INTERVENTIONS:
Drug: Capecitabine — 2000 mg/m2, bid, per os, days 1-14, 4 cycles
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m2 iv day 1, 4 cycles
Drug: Capecitabine — 825 mg/m2, bid, per os, only on days of radiation (Monday through Friday)
  Other Names: Xeloda
  Arms: 4xCapOx
Radiation: Radiotherapy — Pelvic radiotherapy dose: 44 Gy on regional nodes, 50 Gy on primary tumor
  Arms: 4xCapOx
Procedure: Rectal cancer surgery — Laparoscopic or open partial or total mesorectal excision (based on exact tumor location and surgeons discretion)

SUMMARY:
The purpose of this study is to determine whether 4 cycles of neoadjuvant CapOx chemotherapy is more effective than the upfront surgery in patients with intermediate risk CRM"-" mid and upper rectal cancer.

DETAILED DESCRIPTION:
This trial aims to investigate the efficacy of neoadjuvant chemotherapy compared to upfront surgery in intermediate risk rectal cancer patients. This is a prospective multicenter open-label randomized phase III clinical trial. Patients will be randomized using an online randomization system to receive either 4 cycles of neoadjuvant CapOx (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 per os bid days 1-14) chemotherapy and surgery or surgery alone. A stratification will be performed based on N stage, tumor location in the middle or upper rectum and clinical center. Patients with cT3-4aN1-2M0, T4aN0M0 cancer in the upper rectum and сТ2-Т3bN1M0 (based on preoperative MRI) cancer in the middle rectum are included. All patients are potential candidates for adjuvant chemotherapy, according to preoperative staging. Chemoradiotherapy (50 Gy with concomitant capecitabine 825 mg/m2 per os bid on radiation days) will be performed for patients with tumor progression after neoadjuvant chemotherapy. The decision to proceed with adjuvant chemotherapy postoperatively will be based on pTNM stage in both treatment arms, according to actual treatment guidelines. The target accrual is 280 patients in each treatment arm (including 10% potential data loss) based on potential benefit of 10% 3-yr disease-free survival (75% vs 85%), α=0,05, power 80% in the experimental arm. An interim analysis is planned after 50% of the patients will reach a 3-year followup. Pelvic Magnetic Resonance Imaging (MRI) is performed in all patients for staging before and after neoadjuvant chemotherapy and before surgery. Pelvic MRI isbject to central review. Conduction of this study and data collection are controlled by a local institutional board.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically verified colon rectal adenocarcinoma
* cT3-4aN1-2M0 cancer of the upper rectum or сТ2-Т3bN1M0 cancer of the middle rectum (based on pelvic MRI)
* Tumor more than 2 mm from mesorectal fascia (based on pelvic MRI)
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Haemoglobin (HGB) > 90 g/L
* Platelet Count (PLT) > 120x10*9/L
* Serum creatinine < 150 µmol/L
* Total bilirubin < 25 µmol/L

Exclusion Criteria:

* inability to obtain informed consent
* distant metastases
* synchronous or metachronous tumors
* previous chemotherapy or radiotherapy
* clinically significant cardiovascular disorders (myocardial infarction < 6 months before visit, stroke < < 6 months before visit, instable angina < 3 months before visit, arrhythmia, uncontrolled hypertension > 160/100 mm hg
* clinically significant neurological disorders
* previous neuropathy 2 or higher
* current infection or heavy systemic disease
* pregnancy, breastfeeding
* ulcerative colitis
* individual intolerance to treatment components
* proven dihydropyrimidine dehydrogenase (DPD) deficiency
* participation in other clinical trials
* psychiatric disorders, which render patient unable to follow instructions or understand his/her condition
* technical inability to perform pelvic MRI
* inability of long-term followup of the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Adjuvant chemotherapy compliance | 6 months
  Proportion of patients who receive a complete course of adjuvant chemotherapy
Acute chemotherapy toxicity | 14 weeks
  Toxicity measured according to NCI-CTCAE v.5.0
pathologic complete response rate (pCR) | 1 month
local recurrence rate | 3 years
3-year overall survival | 3 years
Operative morbidity | 30 days
  Morbidity measured according to Clavien-Dindo classification
Neoadjuvant chemotherapy disease progression rate | 14 weeks
  Proportion of patients with disease progression during neoadjuvant chemotherapy
Preoperative tumor-associated complications rate | 14 weeks
  The rate of tumor-associated complications (bowel obastruction, bleeding etc) during neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zaman Z Mamedli, PhD, Principal Investigator — N.N.Blokhin Russian Cancer Research Center
Locations (1):
- N.N.Blokhin Russian Cancer Research Center, Moscow, Russia